CLINICAL TRIAL: NCT03167723
Title: Prospective Evaluation of 14F Thal Tube vs 28 French Chest Tube for Hemothorax and Use of Maximum Barrier Precautions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00081328; Pro00020984 (Other: Atrium Health)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-08

CONDITIONS: Hemothorax; Hemopneumothorax; Traumatic; Empyema; Chest Tube Size
Keywords: Chest tube size; Hemothorax; Empyema
MeSH Terms: conditions — Hemothorax; Hemopneumothorax; Empyema

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator masked to outcomes data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 28 French chest tube for hemothorax (Experimental): 28 French straight chest tube placed for non-emergent drainage of hemothorax or hemopneumothorax
  Interventions: Device: Chest tube placement
- 14 French chest tube for hemothorax (Experimental): 14 French thal chest tube placed for non-emergent drainage of hemothorax or hemopneumothorax
  Interventions: Device: Chest tube placement

INTERVENTIONS:
Device: Chest tube placement — Placing tube thoracostomy for hemothorax or hemopneumothorax utilizing maximal barrier precautions.

SUMMARY:
Traumatic hemothorax and hemopneumothorax are common diagnoses which are typically treated by placement of a chest tube. 28-32 Fr chest tubes have previously been shown equivalent to 36-40 Fr chest tubes for the non-emergent drainage of hemothorax. A smaller study has found 14 Fr pigtails had less pain than larger tubes but was not powered to compare outcomes. We seek to perform a prospective randomized trial that is adequately powered comparing efficacy of 14 Fr thal tubes to 28 Fr chest tubes for non-emergent drainage of hemothorax and hemopneumothorax. Additionally, we will employ maximal barrier precautions for all chest tube insertions and compare empyema rates to our historical controls.

ELIGIBILITY:
Inclusion Criteria:

* The patient is admitted to the trauma service.
* The patient has a hemothorax and/or or hemopneumothorax, requiring thoracostomy tube placement.
* Thoracostomy tube placement is able to be performed or witnessed by an investigator listed on the study.
* The patient has not had a chest tube in the past year.
* The patient is >18 years of age.
* In the event the patient is decisionally impaired, consent will be obtained from the individual's legally authorized representative (LAR) or from the individual's healthcare power of attorney (HPA).
* In the instance of reversible impairment, initial consent would be obtained from the LAR/HPA and the patient will be approached for consent once he/she is deemed mentally competent by the care provider.

Exclusion Criteria:

* The patient is incarcerated
* The patient is known to be pregnant
* The patient is < 18 years of age
* The patient is hemodynamically unstable, requiring emergent chest tube placement (in <10 minutes from evaluation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley W Thomas, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karmy-Jones R, Holevar M, Sullivan RJ, Fleisig A, Jurkovich GJ. Residual hemothorax after chest tube placement correlates with increased risk of empyema following traumatic injury. Can Respir J. 2008 Jul-Aug;15(5):255-8. doi: 10.1155/2008/918951. PMID 18716687
- [Result] Inaba K, Lustenberger T, Recinos G, Georgiou C, Velmahos GC, Brown C, Salim A, Demetriades D, Rhee P. Does size matter? A prospective analysis of 28-32 versus 36-40 French chest tube size in trauma. J Trauma Acute Care Surg. 2012 Feb;72(2):422-7. doi: 10.1097/TA.0b013e3182452444. PMID 22327984
- [Result] Kulvatunyou N, Erickson L, Vijayasekaran A, Gries L, Joseph B, Friese RF, O'Keeffe T, Tang AL, Wynne JL, Rhee P. Randomized clinical trial of pigtail catheter versus chest tube in injured patients with uncomplicated traumatic pneumothorax. Br J Surg. 2014 Jan;101(2):17-22. doi: 10.1002/bjs.9377. PMID 24375295
- [Derived] McCartt J, Ross SW, Cunningham KW, Wang H, Sealey L, Brake J, Christmas A, Sachdev G, Green J, Thomas BW. A Randomized Non-Inferiority Clinical Trial of 14Fr Thal versus 28Fr Tube Thoracostomy for Traumatic Hemothorax. Am Surg. 2025 Apr;91(4):579-586. doi: 10.1177/00031348241308907. Epub 2024 Dec 19. PMID 39700058

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n=84) Hemodynamic instability (n=36) Chest tube placed at outside facility (n=12) Multiple chest tube placement (n=10) Declined to participate (n=1) Not meet inclusion criteria (n=6) Other reasons (n=19)
Period: Overall Study
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Started | 55 | 54
Completed | 51 | 48
Not Completed | 4 | 6
Not completed — Protocol Violation | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49.9 [33.6 to 72.4] | 46.5 [26.8 to 68.6] | 49 [26.5 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 38 | 39 | 77
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Injury Severity Score - score that ranges from 3 (least) to 75 (most) injured [Median (Inter-Quartile Range); unit: units on a scale] — Specific injuries in each body region are coded on a scale of 1 (minor), 2 (moderate), 3 (serious, not life threatening), 4 (severe, life threatening, survival probable), 5 (critical, survival uncertain) and 6 (unsurvivable).
  units on a scale | 17 [13 to 29] | 18 [10 to 29] | 17 [10 to 29]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Retained Hemothorax Following Initial Chest Tube Placement Requiring Intervention
Description: Number of Participants with Retained hemothorax requiring an additional intervention, either video-assisted thoracoscopic surgery (VATS) or additional thoracostomy tube placement.
Time Frame: 90 days
Measure: Number; unit: Number of Participants
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
Number of Participants | 51 | 48
Statistical Analysis 1: Comparison: 28 French Chest Tube for Hemothorax vs 14 French Chest Tube for Hemothorax; Test type: Non-Inferiority — 15% Non-Inferiority; p = 0.036, Farrington-Manning

2. Secondary Outcome: Duration of Chest Tube Placement.
Description: Number of days with chest tube placement
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
days | 3.9 [2.6 to 5.3] | 3.9 [2.8 to 5.8]

3. Secondary Outcome: Number of Participants Stratified by Length of Hospitalization Stay
Description: Number of weeks spent in hospital
Time Frame: 90 days
Measure: Number; unit: Number of Participants
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
Number of Participants
  1 Week | 20 | 15
  2 Weeks | 19 | 15
  3 Weeks | 7 | 6
  > or = 4 Weeks | 5 | 12

4. Secondary Outcome: Change in Subjective Pain Scores From Baseline at 90 Days
Description: Assessed with 0-10 numeric pain rating scale - the higher the number, the more severe the pain
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
units on a scale | 0 [-1 to 2] | 0 [-2 to 2]

5. Secondary Outcome: Hemodynamic Stability Post-insertion
Description: determined by vital signs: temperature, heart rate, blood pressure, oxygen saturation (Systolic Blood Pressure <90mm Hg)
Time Frame: 90 days
Measure: Number; unit: Number of Participants
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
Number of Participants | 2 | 1

6. Secondary Outcome: Initial Drainage From Chest Tube at 5 Minutes
Description: Milliliters of chest tube drainage at 5 minutes
Time Frame: 5 Minutes
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
mL | 150 [60 to 500] | 100 [3.5 to 350]

7. Secondary Outcome: Tube Specific Complications: Air Leak, Tube Malposition, & Tube Migration
Description: Number of Tube specific complications: Air leak, tube malposition, & tube migration
Time Frame: 90 days
Measure: Number; unit: Ocurrences
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
Ocurrences | 7 | 5

8. Secondary Outcome: Time to Radiographic Resolution of Pneumothorax/Hemothorax/Hemopneumothorax
Description: Number of days until radiographic resolution of pneumothorax/hemothorax/hemopneumothorax
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
days | 0.5 [0.1 to 2.7] | 1 [0.1 to 2.7]

9. Secondary Outcome: Recurrent Pneumothorax/Hemothorax/Hemopneumothorax After Tube Removal
Description: Number of Participants with Recurrent pneumothorax/hemothorax/hemopneumothorax after tube removal
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
participants | 5 | 1

10. Secondary Outcome: Readmission for Chest Tube Related Complications
Description: Number of Participants readmitted for chest tube related complications
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
Number analyzed (Participants) | 51 | 48
participants | 9 | 4

ADVERSE EVENTS:
Time Frame: 90 days
Description: Participants will be monitored for serious adverse events from the moment of randomization through 90 days post tube insertion. Due to their mechanism of injury and high trauma burden, participants are expected to have significant trauma related complications. AEs or SAEs determined to be unrelated to study procedure or tube size will not be reported to the IRB. Submission of any serious adverse event will not occur until relatedness of the event has been determined.
Arm/Group | 28 French Chest Tube for Hemothorax | 14 French Chest Tube for Hemothorax
All-Cause Mortality (participants affected / at risk) | 2/55 | 2/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT03167723/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03167723/ICF_001.pdf